CLINICAL TRIAL: NCT04386239
Title: Pilot Study on the Use of Sarilumab in Patients With COVID-19 Infection
Brief Title: Study on the Use of Sarilumab in Patients With COVID-19 Infection
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Technical impasse from IRB
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Stefano Rusconi, Co-investigator, ASST Fatebenefratelli Sacco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-SARI-001
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: COVID19
Keywords: Coronavirus; Pandemic; Lombardy
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sarilumab

STUDY DESIGN:
Intervention Model Description: Monocentric, escalation dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Covid-19 (Experimental): Patients with documented (chest X-Ray or Computed Tomography scan) Covid-19 (Polymerase Chain Reaction+ swab test) interstitial pneumonia and BCRSS ≥3 and <4 will be requested consent to the study.
  Interventions: Drug: Sarilumab Prefilled Syringe

INTERVENTIONS:
Drug: Sarilumab Prefilled Syringe — Sarilumab administration must be associated with an antiviral treatment as defined by the treatment protocol suggested by the SIMET Experts group 4 and AIFA recommendations: chloroquine 500 mg 1 tablet twice daily or hydroxychloroquine 400 mg 1 tablet twice daily in the first day and then 200 mg 1 tablet twice daily.
  Other Names: Sarilumab

SUMMARY:
Sarilumab is an anti-interleukin-6 human monoclonal antibody, such as tocilizumab, which is administered subcutaneously every two weeks for the treatment of moderate to severe active rheumatoid arthritis in adult patients. Despite the effectiveness reported for tocilizumab in the recently published experiences, the need to rapidly find alternative therapies to manage the complications of Covid-19 infection remains extremely high. The lack of clinical experience on the usage of sarilumab in such patients prevents the possibility of adopting early access programs for using commercially available sarilumab (prefilled syringe) packs in patients with severe Covid-19 pneumonia. The present study is aimed to generate a rapid, still robustly documented, evidence on the potential clinical efficacy and tolerability of a further IL-6R antagonist in Covid-19 pneumonia.

DETAILED DESCRIPTION:
In February 2020, the emergence of the COVID-19 epidemic in Italy and, especially, in Lombardy, with a potential fatal outcome in a significant proportion of cases, determined the need for adopting new therapeutic approached based on the few data available in literature. Although there are no clinical data available in COVID-19 patients concomitantly treated with Sarilumab subcutaneously (SC) nor intravenously (IV), there is scientific rationale that supports the exploration of sarilumab to treat pulmonary complications related to Covid-195-6. By inhibiting interleukin-6 (IL-6)signaling, sarilumab may potentially interrupt cytokine-mediated pulmonary injury precipitated by infection with SARS-CoV-2 and thereby ameliorate severity and/or reduce mortality among patients presenting with Covid-19 pneumonia when administered in conjunction with antiviral therapy. given the apparent dose/dose pharmacokinetic/ pharmacodynamic (PK/PD) equivalence of 400 mg of tocilizumab to 400 mg of sarilumab, we propose a dose escalation protocol by which the first 5 included patients will be treated with a dosage of 200 mg of sarilumab IV as 1st dose, followed by clinical reassessment after 12 hours and in case of no major adverse events and lack of improvement in respiratory function and / or persistence of fever and persistently high inflammatory markers re-administration of 200 mg intravenous (IV) of sarilumab. If no patients showed unfavorable safety signals, and no clear improvement is detected in >50% of the initially treated five patients after 96 hours since last administration, the dosage will be increase to sarilumab 400 mg IV as first and second dose in the remaining patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 85 years.
* Documented (chest X-Ray or TC scan), severe (BCRSS ≥3 and <4) interstitial pneumonia with respiratory failure (requiring supplemental oxygen) with positive Covid-19 swab testing.
* Worsening of respiratory exchanges such as to require ventilation with Venturi mask >31% (6L/minute).
* Increased levels of D-dimer (> 1500 ng/mL) or D-dimer progressively increasing (over 3 consecutive measurements) and reaching ≥ 1000 ng/mL.
* Signed informed consent.

Exclusion Criteria:

* Age < 18 years or ≥ 85 years.
* AST / ALT > 5x Upper normal limit.
* Neutrophil count lower than 500 cells / mL.
* Platelet count lower than 50,000 cells / mL.
* Documented sepsis due to infections other than Covid-19.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who show an improvement of the respiratory function | 6 weeks
  Clinical efficacy of sarilumab in adult patients hospitalized due to severe Covid-19 pneumonia based on the proportion of patients who show an improvement of the respiratory function, described as ≥30% decrease in oxygen requirement compared to baseline (as defined as the ratio of O2 flow through the Venturi mask).

SECONDARY OUTCOMES:
Evaluation of the time to resolution of fever | 6 weeks
  Evaluation of the time to resolution of fever, defined as body temperature ≤36.6°C axilla, ≤37.8°C rectal or tympanic for at least 48 hours without antipyretics in patients with fever at baseline.
Evaluation of the viral load on blood and sputum for COVID-19 | Before administration of sarilumab, 48 hours and 96 hours after administration
  Evaluation of the viral load on blood and sputum for COVID-19
Evaluation of the plasma concentration of GM-CSF | Pre-treatment and 96 and 120 hours post-treatment
  Evaluation of the plasma concentration of GM-CSF
Evaluation of the plasma concentration of Il-6 | Pre-treatment and 96 and 120 hours post-treatment
  Evaluation of the plasma concentration of Il-6
Evaluation of the plasma concentration of TNF-α | Pre-treatment and 96 and 120 hours post-treatment
  Evaluation of the plasma concentration of TNF-α
Evaluation of the rate of progression of White Blood Cell (WBC) fraction | 96 and 120 hours post-treatment
  Evaluation of the rate of progression of WBC fraction of immature granulocytes - IG - (absolute count).

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Galli, Professor, Principal Investigator — University of Milan
Locations (1):
- Divisione Clinicizzata di Malattie Infettive, ASST FBF-Sacco, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04386239/Prot_SAP_000.pdf